CLINICAL TRIAL: NCT00851383
Title: A Phase I Placebo-controlled, Double-blinded (in Terms of Vaccine or Placebo), Randomized Dose-escalation Trial to Evaluate the Safety and Immunogenicity of Ad35-GRIN/ENV HIV Vaccine in Healthy Adult Volunteers. (IAVI B001)
Brief Title: A Trial to Evaluate Ad35-GRIN/ENV HIV Vaccine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI B001
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Human Immunodeficiency Virus; HIV Seronegativity; Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): Ad35-GRIN/ENV: 2x10^9 vp
  Interventions: Biological: Ad35-GRIN/ENV
- Group B (Experimental): Ad35-GRIN/ENV: 2x10^10 vp
  Interventions: Biological: Ad35-GRIN/ENV
- Group C (Experimental): Ad35-GRIN/ENV: 2x10^11 vp
  Interventions: Biological: Ad35-GRIN/ENV
- Group D (Experimental): Ad35-GRIN at 1x10^10 vp
  Interventions: Biological: Ad35-GRIN

INTERVENTIONS:
Biological: Ad35-GRIN/ENV — This is a dose-escalation trial. Each group will receive the Ad35-GRIN/ENV vaccine at different dosage levels.
  Arms: Group A; Group B; Group C
Biological: Ad35-GRIN — This is a dose-escalation trial. Group D will receive the Ad35-GRIN vaccine.
  Arms: Group D

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of Ad35-GRIN/ENV HIV vaccine and Ad35-GRIN HIV vaccine administered intramuscularly at 0 and 6 months.

DETAILED DESCRIPTION:
This study is a phase I dose-escalation randomized, placebo-controlled study designed to evaluate the safety and immunogenicity of Ad35-GRIN and Ad35-ENV filled in the same vial and administered as a single, combined vaccine. This is the first administration of this vaccine in humans. The study will be double blind with respect to vaccine or placebo. The vaccine will be administered intramuscularly at months 0 and 6 at three dose levels: 2 x 10^9, 2 x 10^10, and 2 x 10^11 vp per dose. Volunteers will be randomized to vaccine: placebo in a 10:4 ratio in each group. A fourth group was added as a protocol amendment to study Ad35-GRIN HIV vaccine alone at 1x10^10 vp in 14 volunteers (10:4 vaccine:placebo).

Volunteers will be screened up to 42 days before vaccination (90 days for Ad35 neutralizing antibody screening) and will be followed for 12 months after the last vaccination (18 months total study participation). Estimated enrollment will take approximately 5 months. Thus, the total duration of the study would be approximately 23 months.

ELIGIBILITY:
Inclusion Criteria

* Healthy males and females, as assessed by a medical history, physical exam, and laboratory tests
* Willing to comply with the protocol and follow up for the planned duration of the study (screening plus 18 months)
* In the opinion of the PI or designee, has understood the information provided. Written informed consent needs to be given before any study-related procedures are performed
* Amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required visit, and willing to continue 5 yrs of annual follow-up contact
* Demonstrates understanding (assessment of understanding will be performed) of the risk for harm observed in the STEP Study results
* Assessed by the clinic staff as being at "low risk" for HIV infection on the basis of sexual behaviors within the 12 months prior to enrolment defined as follows:
* Sexually abstinent OR
* Had two or fewer mutually monogamous relationships with partners believed to be HIV-uninfected and who did not use illicit drugs ( methamphetamines (crystal meth), heroin, cocaine, including crack cocaine or chronic marijuana abuse) OR
* Had two or fewer partners believed to be HIV-uninfected and who did not use illicit drugs (methamphetamines (crystal meth), heroin, cocaine, including crack cocaine or chronic marijuana abuse), and with whom he/she regularly used condoms for vaginal and anal intercourse
* Willing to undergo HIV Testing, HIV counseling and receive HIV Test results
* If sexually active female, using an effective method of contraception (hormonal contraceptive; diaphragm; Intra Uterine Device (IUD); condoms; anatomical sterility in self or partner) from screening until at least 4 months after last vaccination. All female volunteers must be willing to undergo urine pregnancy tests at time points as indicated in the Schedule of Procedures
* If sexually active male, willing to use an effective method of contraception (such as condoms, anatomical sterility) from screening until 4 months after the last vaccination

Exclusion Criteria

* Confirmed HIV-1 or HIV-2 infection
* Detection of Ad35-specific serum neutralizing antibody
* Reported high-risk behavior for HIV infection defined as:

  * Within 12 months before vaccination, the volunteer has:
  * Had unprotected vaginal or anal sex with a known HIV infected person or a casual partner (i.e. no continuing established relationship)
  * Engaged in sex work for money or drugs.
  * Excessive daily alcohol use or frequent binge drinking or chronic marijuana use or use of other illicit drugs.
  * Recently acquired a sexually transmitted disease (STD) including syphilis, gonorrhoea, non-gonococcal urethritis, Trichomonas vaginalis, symptomatic Herpes genitalis (HSV-2), chlamydia, pelvic inflammatory disease (PID), mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B).
  * Has a high-risk partner either currently or had such a partner within the previous 12 months.
* Any clinically significant abnormality on history or examination, including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical steroids and inhaled steroids for sinus decongestion are permitted), immunosuppressive, antiviral, anticancer, anti-tuberculosis, or other medications considered significant by the investigator within the previous 6 months;
* Any clinically significant acute or chronic medical condition that is considered progressive or, in the opinion of the investigator, would make the volunteer unsuitable for the study.

Any of the following abnormal laboratory parameters

* Hemoglobin <11.0 g/dL for women and <12.5 g/dL for men
* Absolute Neutrophil Count (ANL): ≤ 999/mm3
* Absolute Lymphocyte Count (ALC): ≤ 500/mm3
* Platelets: ≤ 90,000 ≥ 550,000/mm3
* Creatinine: >1.1 ULN
* AST: >1.25 x ULN
* ALT: >1.25 x ULN
* Urinalysis 2+ by urine dipstick

  * Blood (not due to menses);
  * Protein
  * Leucocytes
* Confirmed diagnosis of hepatitis B (surface antigen HbsAg), hepatitis C (HCV antibodies), or active syphilis
* If female, pregnant or planning a pregnancy within 4 months after last vaccination; or lactating
* Receipt of live attenuated vaccine within the previous 60 days (live attenuated flu vaccine within 14 days) or planned receipt within 60 days after vaccination with Investigational Product or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product
* Receipt of blood transfusion or blood products within the previous 6 months
* Participation in another clinical study of an investigational product currently, within the previous 3 months or expected participation during this study
* Receipt of another investigational HIV vaccine candidate at any time
* History of severe or very severe local or systemic reactogenicity to vaccines or history of severe allergic reactions
* Major psychiatric illness, including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, suicidal attempt or ideation in the previous 3 yrs
* Unwilling to forgo donations of blood, sperm, eggs, bone marrow or organs during the study
* Asplenia: any condition resulting in the absence of a spleen

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity signs and symptoms, laboratory measures, and adverse events) | 18 months

SECONDARY OUTCOMES:
Immunogenicity: Proportion of volunteers with HIV-1 specific T-cell responses by ELISPOT assay. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keefer, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Keefer MC, Gilmour J, Hayes P, Gill D, Kopycinski J, Cheeseman H, Cashin-Cox M, Naarding M, Clark L, Fernandez N, Bunce CA, Hay CM, Welsh S, Komaroff W, Hachaambwa L, Tarragona-Fiol T, Sayeed E, Zachariah D, Ackland J, Loughran K, Barin B, Cormier E, Cox JH, Fast P, Excler JL. A phase I double blind, placebo-controlled, randomized study of a multigenic HIV-1 adenovirus subtype 35 vector vaccine in healthy uninfected adults. PLoS One. 2012;7(8):e41936. doi: 10.1371/journal.pone.0041936. Epub 2012 Aug 3. PMID 22870265
- See also: International AIDS Vaccine Initiative — http://www.iavi.org